CLINICAL TRIAL: NCT02538432
Title: 15xxGCC: PHASE II TRIAL OF THE EP4 RECEPTOR ANTAGONIST, AAT-007 (RQ-07; CJ-023,423) IN ADVANCED SOLID TUMORS
Brief Title: Phase II Trial of EP4 Receptor Antagonist, AAT-007 (RQ-07; CJ-023,423) in Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI No Longer at University of Maryland. Now at Fox Chase
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15XXGCC
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer; Non-Small Cell Lung Cancer; Breast Cancer
Keywords: Disease Progression; Non-Responsive Disease; Advanced Disease
MeSH Terms: conditions — Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Disease Progression | interventions — grapiprant; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RQ-00000007 Alone (Experimental): RQ-0000007 250 mg will be self-administered orally, with or without food, each morning and evening, approximately 12 hours apart.
  Interventions: Drug: RQ-00000007
- Gemcitabine (Active Comparator): For patients with breast or lung cancer who have not previously received gemcitabine as part of their therapy or who may benefit from re-challenge with gemcitabine, gemcitabine will be given as an IV.
  Interventions: Drug: RQ-00000007; Drug: Gemcitabine

INTERVENTIONS:
Drug: RQ-00000007 — RQ-07 250 mg will taken orally, with or without food, each morning and evening, approximately 12 hours apart. Drug administration will be continuous. Every 21 day period will be considered one cycle of treatment.
  Other Names: AAT-007; RQ-07; CJ-023,423
Drug: Gemcitabine — For patients with breast or lung cancer who have not previously received gemcitabine as part of their therapy or who may benefit from re-challenge with gemcitabine, gemcitabine will be administered at 1000 mg/m2 IV over 30 minutes for 3 out of 4 weeks after appropriate pre-medications. Every 4 week period (28 days) will be considered one cycle.
  Other Names: Gemzar
  Arms: Gemcitabine

SUMMARY:
This is a phase II trial of (RQ-07) in advanced solid tumors in prostate, breast or non-small cell lung cancer.

DETAILED DESCRIPTION:
This is a phase II trial of (RQ-07) in advanced solid tumors in advanced prostate, breast or lung cancer. The purpose of this trial is to determine whether the administration of the study drug RQ-07 can decrease circulating tumor cells in advanced prostate, breast or lung cancer. Additionally, the study will evaluate whether the study drug may improve outcome in advanced prostate, breast or lungs cancer either by itself or when combined with gemcitabine, a standard chemotherapy drug. The combination of with gemcitabine will only be investigated after disease has worsened with the study drug RQ-07 by itself and only in patients with prostate or lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed breast, prostate or non-small cell lung cancer or other A tissue block, 10 unstained slides or fresh tissue biopsy is required.
2. At least 2 weeks should have elapsed since the last treatment and patients should have recovered from previous significant toxicity (i.e. to grade 1 or less).
3. ECOG Performance Status <2.
4. Patient at least 18 years of age or older.
5. Adequate hematological function as defined by the protocol, section 4.1.5.
6. Patients must have a serum creatinine within normal limits, or an estimated or measured creatinine clearance > 35 mg/ml/min.
7. Normal serum electrolytes (no >grade 2 abnormalities), magnesium and phosphorus on the day of therapy. Correction of abnormalities is permitted.

   Adequate hepatic function per institutional standards (see exclusion).
8. All patients must be informed of the investigational nature of this study and must sign and give written informed consent.
9. Serum calcium, magnesium and potassium must be within normal limits. Supplementation to achieve normal values is permitted.
10. Patients who are potentially fertile and sexually active must be willing to utilize effective birth control.
11. Patients with CNS metastases which are/were symptomatic must have completed therapy (surgery, gamma knife, XRT) and be neurologically stable.
12. Patients must have > or = 4 circulating tumor cells

Exclusion Criteria:

1. Patients must not have serious infection or other serious underlying medical condition which would impair the ability of the patient to receive protocol treatment.
2. Current uncontrolled cardiac disease
3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
4. Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 4 weeks of registration.
5. Patients with acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition or patients known to be HIV positive
6. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Circulating Tumor Cells (CTC) | Day 21
  The efficacy of the treatment drug will be assessed by the reduction of the number of CTCs. Blood sample collection will be done to assess CTCs.

SECONDARY OUTCOMES:
Myeloid Derived Suppressor Cell (MDSC) | Day 21
  The efficacy of the treatment drug RQ-07 will be assessed as a single agent and in combination with gemcitabine in breast cancer and lung cancer patients only. MDSC evaluation will be done via a blood sample collection

CONTACTS AND LOCATIONS:
Overall Officials: Martin Edelman, M.D., FACP, Principal Investigator — University of Maryland Greenebaum Cancer Center

IPD SHARING:
Plan to Share IPD: No